CLINICAL TRIAL: NCT06156254
Title: Impact of a Community Care Intervention to Address Inequities in COVID-19 and Influenza Vaccination Among Adults Suffering From Disproportionate Chronic Disease
Brief Title: Community Care Intervention to Decrease COVID-19 Vaccination Inequities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Clinical Directors Network (Network); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HCAAD148; R01MD017232 (NIH)
Record Dates: First submitted 2023-11-29; First posted 2023-12-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Vaccination

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker (CHW) Intervention to Enhance Vaccination Behavior (Experimental): Patients randomized to the CHW intervention will receive up to 3 psychoeducational sessions in English or Spanish targeting the specific reason(s) why a patient is not up to date with their COVID-19 vaccine. CHWs will use motivational interviewing techniques to promote vaccination behaviors.
  Interventions: Behavioral: Community Health Worker Intervention to Enhance Vaccination Behavior (CHW-VB)
- Usual Care (No Intervention): Patients will receive the care that they would usually receive independent of the study but won't have access to the intervention.

INTERVENTIONS:
Behavioral: Community Health Worker Intervention to Enhance Vaccination Behavior (CHW-VB) — Patients randomized to the CHW intervention will receive up to 3 psychoeducational sessions in English or Spanish targeting the specific reason(s) why a patient is not up to date with their COVID-19 vaccine. CHWs will use motivational interviewing techniques to promote vaccination behaviors.
  Arms: Community Health Worker (CHW) Intervention to Enhance Vaccination Behavior

SUMMARY:
The purpose of this study is to find out if a community health workers (CHW) intervention conducted in Federally Qualified Health Centers (FQHCs) can increase the number of adults with chronic illnesses who are up-to-date with their COVID-19 and influenza vaccines.

DETAILED DESCRIPTION:
Many factors contribute to inequities in vaccination rates among racial and ethnic minorities, including differences in vaccine acceptance and intention and related variability in social behavioral norms, knowledge, risk perception, trust, and structural barriers. The World Health Organization has called for community health workers (CHWs) as a key strategy to address vaccination inequities among vulnerable populations worldwide. CHWs are trusted messengers and cultural brokers that can address barriers to vaccination access and provide language, culturally, and literacy-appropriate information to promote awareness of and motivation to partake in protective vaccination behaviors. CHWs can have a central role in Federally Qualified Health Centers (FQHCs) by helping link their mostly non-White patients with health care and community resources.

This study examines whether a CHW intervention can be effective in increasing vaccination rates by providing education, help with behavior changes, and assistance in navigating barriers to increase equal access to vaccination. The CHW intervention consists of up to 3 psychoeducational sessions in English or Spanish targeting the specific reason(s) why a patient is not up to date with their COVID-19 vaccine. According to the reason(s), the CHW implements strategies to educate, motivate, and help navigate any access barriers to getting vaccinated. CHWs use motivational interviewing techniques to encourage patients to get vaccinated. Patients also receive educational flyers designed by a local artist addressing their own COVID-19 vaccination knowledge gaps. Toward the end of each session, the CHW works with the patient to create a Patient Action Plan with steps the patient can take to overcome their barriers to vaccination.

RAND and Clinical Directors Network (CDN) are conducting a randomized controlled trial (RCT) in New York City FHQCs to determine the efficacy of the CHW intervention to improve vaccine acceptance and uptake among racial/ethnic minority adults with any of 7 chronic conditions (asthma, diabetes, hypertension, obesity, depression, anxiety disorder, or PTSD). This research study plans to randomly assign (like the flip of a coin) a total of 800 patients to a "Usual Care Group" (400 patients who will continue to receive usual care with no changes) or "CHW Group" (400 patients who will receive the CHW intervention and usual care).

The following four research questions guide the study:

* What makes being up to date for COVID and Flu vaccines difficult for people with chronic illness?
* Can a CHW intervention help patients be up to date with the COVID and Flu vaccines?
* What about the CHW intervention specifically works for different types of patients?
* What can help expand the CHW program to more people for a longer time?

The main study hypothesis is that participants assigned to the intervention will exhibit significantly higher vaccine acceptance and actual increases in vaccination rates.

If the intervention is effective, it has the potential to decrease disparities in severe illness resulting from COVID-19 and influenza by increasing vaccination rates among racial and ethnic minority populations with chronic illness. Since FQHCs employ CHWs to help deliver care to patients with chronic illnesses, the intervention would be easily implementable and scalable for future COVID-19 and influenza vaccination seasons.

ELIGIBILITY:
Inclusion Criteria:18 years or older AND speak English or Spanish AND have no obvious physical or cognitive impairment that would make them unable to complete the assessment (as indicated by confusion or inability to understand the questions).

Exclusion Criteria: not willing to consent OR acutely sick OR have high suicide risk

Eligibility criteria: Have received a COVID-19 vaccine but not received an updated COVID-19 vaccine at the time of recruitment AND self-report being told by a physician they have one of the following health conditions; high blood pressure/hypertension OR diabetes OR asthma OR overweight/obese OR a one of the following mental health condition (probable depression, probable generalized anxiety, or probable PTSD)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccine acceptance | Baseline and 3 months
  COVID-19 vaccine acceptance at 3 months is measured by a survey self-report survey item asking participants to rate the following statement on a 5-to Likert scale (from 1 = strongly disagree to 5 = strongly agree): "If I was not up-to-date with the COVID-19 vaccines recommended for me, I would get the missing vaccinations." This variable is dichotomized to COVID-19 vaccine acceptance (0 = strongly disagree/disagree/neutral; 1 = agree/strongly agree)
COVID-19 vaccine uptake | Baseline and 3 months
  COVID-19 vaccine uptake is defined based on information gathered by multiple sources combining data obtained from patient survey self-reports, EHR data, and Healthix data. We also confirm receipt of the vaccine by asking the participant to see their COVID-19 vaccination card. Vaccination extracted data is from Healthix, the largest Regional Health Information Organization (RHIO) and from a wide array of facilities providing vaccinations will be pulled, including hospitals, health centers, ambulatory care sites, community vaccination sites, and pharmacies.

SECONDARY OUTCOMES:
Influenza vaccine uptake | Baseline and 3 months
  As for COVID-19 update, we rely on a combination of survey self-report, EHR, and Healthix data.

CONTACTS AND LOCATIONS:
Overall Officials: Marielena Lara, MD, MPH, Principal Investigator — RAND; Lisa Meredith, PhD, Principal Investigator — RAND; Jonathan Tobin, PhD, Principal Investigator — Clinical Directors Network; Andrea Cassells, MPH, Study Director — Clinical Directors Network
Locations (4):
- United States (4):
  - Brownsville Multi-Service Health Center, Brooklyn, New York
  - Bedford-Stuyvesant Family Health Center, Brooklyn, New York
  - Community Healthcare Network, New York, New York
  - Morris Heights Health Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
We will deposit deidentified participant-level data, survey instruments, and variable descriptions to the NIMH Data Archive in accordance with the NIH Data Management and Sharing Policy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available by the completion of the study on 2/28/27
Access Criteria: The study's deidentified participant-level data will be made publicly available

REFERENCES:
- [Derived] Meredith LS, Tobin JN, Cassells A, Howell K, Hernandez HG, Gidengil C, Williamson S, Dong L, Timmins G, Alvarado G, Holder T, Cortez Lainez J, Lin TJ, Lara M. Boost your health (Refuerza tu Salud): Design of a randomized controlled trial of a community health worker intervention to reduce inequities in COVID-19 and influenza vaccinations. Contemp Clin Trials. 2025 Jun;153:107848. doi: 10.1016/j.cct.2025.107848. Epub 2025 Feb 16. PMID 39965727